CLINICAL TRIAL: NCT01633021
Title: Development of the Family Map: Examination of Communal Coping Across Disease Context
Brief Title: Developing the Family Map: Looking at Communal Coping
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912149; 12-HG-N149
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: Sickle Cell; Diabetes; Cancer; Cardiovascular Disease; Genetic Screening
Keywords: Support; Cancer; Network; Diabetes; Sickle Cell Trait / Sickle Cell Disease; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Cardiovascular Diseases; Sickle Cell Trait; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes: Self/Family member affected by type-2 diabetes (plus self-referred family-members)
- Heritable Cancer Screen-Positive: Person who has screened-positive for heritable cancers on genetic tests (plus referred family-members)
- Sickle Cell (Trait/Disease/Related): Self/Family member affected by Sickle Cell Trait or Sickle Cell Disease (plus self-referred family-members)

SUMMARY:
Background:

- Knowing one s family medical history is a part of staying healthy. Some health risks run in families, and knowing these risks can promote more healthy behavior. Different social and cultural factors may affect how family members share this information. Genetic risk information that is shared in one family may not be shared in the same way in another. This information may also be shared differently between spouses, siblings, or parents and children. It may even be shared with more distant relatives. Knowing the information that family members share and how they share it may help researchers improve genetic disease treatment and support plans. Family surveys of people who have genetic health risks may help provide this information.

Objectives:

- To study how family members affected by genetic-related diseases share health information with each other.

Eligibility:

* Individuals at least 18 years of age who can read English or Spanish.
* Participants affected by a genetic disease or be related or married to someone who has the disease.

Design:

* Participants will be screened with an initial questionnaire. They will identify their genetic disease and provide a basic health history.
* Participants who have the disease will complete an online survey or participate in a personal interview. The questions will take about 45 minutes to 1 hour to answer. The survey will ask about family health history and family support. Participants will also provide referrals to a spouse or relatives who will participate in the study.
* The spouse or relative will answer a similar survey. The survey will ask about health history and support for the spouse/relative with the disease.
* A gift card will be given as thanks for participating in the study.

DETAILED DESCRIPTION:
Facilitating the dissemination of disease risk information and promoting engagement in healthful behaviors within families may be enhanced by using network-based interventions. Network-based interventions are innovative in that they are tailored to the structure of the social system within which individuals are embedded. Understanding the social and relational factors associated with processes of family risk dissemination, family encouragement, and support is essential to developing network-based intervention tools targeting the family. The first objective of the current project is to ascertain those key social pathways that can be used in a family-centered network-based intervention that promotes disease prevention and health promotion in at-risk families. To this end, efforts will be focused on assessing whether there is a consistent, small set of relational characteristics associated with the dissemination of family risk information and processes of both behavioral and emotional adaptation to disease risk across various disease and cultural contexts. The second objective is to examine the feasibility of using cognitive network approaches to assess social interactions among family members as a means to enhance the implementation of a network-based intervention. A cognitive network is an individual's perception of the relationships among their family (or network) members. Thus, cognitive network approaches can potentially be used to capture an accurate representation of family social structure based on the information provided by a small subset of optimally situated family members. Those key social pathways identified within the first objective of this research will be used to address the second objective. Families affected by diseases and disorders that span the spectrum of genetic penetrance, ranging from highly penetrant, monogenetic disease to less penetrant, common complex conditions, will be recruited for the study. Further, the current effort will seek to engage samples from diverse cultural backgrounds to address our limited knowledge regarding risk communication and adaptation in such families and to facilitate generalization of results. Study participants will be recruited from established cohorts, outreach events, or ongoing studies, both at the NIH and at extramural institutions. Family members will be recruited using a snowball sampling approach and will be asked to complete an in-person, web-based and/or telephone survey/interview. Interviews will have a semi-structured format to allow for slight deviations in prompts and probes to address participant questions. The research addressed in this protocol will lead to the development of an innovative methodology with the potential to improve the design and implementation of family-based interventions that promote disease prevention.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 years or older
* Ability to complete in-person, web-based or telephone survey/interview(s)
* Ability to read English or Spanish (in some cases)
* Affected by or have at least one first- or second-degree relative affected by or have a spouse/partner affected by the disease(s) of interest OR Biological or non-biological (e.g. adopted, step, spouse, family through marriage) relative of the primary participant.

EXCLUSION CRITERIA:

Individuals with cognitive difficulties will be excluded from the study, as participants will be required to comprehend and legally consent to participation in this study and complete the survey/interview(s).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment is appropriate to the disease/screening-specific context, and may work with advocacy groups. Prospective participants who have / are at risk for chronic genetic disease (or are related to someone affected by condition) may be eligible to participate.@@@
Sampling Method: Non-Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2012-07-05 (Actual)

PRIMARY OUTCOMES:
Social & relational factors from family network data | Varies by sub-study
  Identify social and relational factors used to characterize family environment re communication of health information, encouragement of health behaviors, provision of support.

SECONDARY OUTCOMES:
Cognitive network utility evaluation | Varies by sub-study
  Evaluate the utility of cognitive network approaches to characterize the family social environment

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (3):
- United States (3):
  - National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Geisinger Autism & Developmental Medicine Institute, Lewisburg, Pennsylvania

REFERENCES:
- [Background] Lewis MA, McBride CM, Pollak KI, Puleo E, Butterfield RM, Emmons KM. Understanding health behavior change among couples: an interdependence and communal coping approach. Soc Sci Med. 2006 Mar;62(6):1369-80. doi: 10.1016/j.socscimed.2005.08.006. Epub 2005 Sep 16. PMID 16146666
- [Background] Stokols D. Establishing and maintaining healthy environments. Toward a social ecology of health promotion. Am Psychol. 1992 Jan;47(1):6-22. doi: 10.1037//0003-066x.47.1.6. PMID 1539925
- [Background] Ersig AL, Williams JK, Hadley DW, Koehly LM. Communication, encouragement, and cancer screening in families with and without mutations for hereditary nonpolyposis colorectal cancer: a pilot study. Genet Med. 2009 Oct;11(10):728-34. doi: 10.1097/GIM.0b013e3181b3f42d. PMID 19707152
- [Derived] Desine S, Eskin L, Bonham VL, Koehly LM. Social support networks of adults with sickle cell disease. J Genet Couns. 2021 Oct;30(5):1418-1427. doi: 10.1002/jgc4.1410. Epub 2021 Apr 12. PMID 33847032